CLINICAL TRIAL: NCT05422014
Title: Life Care Specialist (LCS) - Pain Management and Prevention of Substance Misuse in Upper Extremity Trauma
Brief Title: Upper Extremity Life Care Specialist (LCS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: American Society for Surgery of the Hand (Other); Ruth Jackson Orthopaedic Society (Unknown)
Responsible Party: Principal Investigator, Nicole Zelenski, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00004303
Record Dates: First submitted 2022-05-24; First posted 2022-06-16 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Upper Extremity Trauma
Keywords: Opioids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LCS Intervention (Experimental): With Opioid Risk Education, patients will receive opioid education after completing the validated Opioid Risk Tool (ORT), a detailed substance abuse survey and mental health screening, and Naloxone education. Therapeutic Intervention will include the Community Resiliency Model CRM), progressive muscle relaxation, sound therapy. Clinical Pain Coordination will include directed referrals for complex needs, including mental health and substance use disorders, as needed. In addition to above mentioned 3 intervention components, all patients in the LCS intervention arm will also receive the current standard-of-care.
  Interventions: Behavioral: Life Care Specialist (LCS)
- No LCS Intervention (No Intervention): Patients will receive the current standard-of-care for pain management in the aftermath of trauma, which includes: a standardized prescription protocol, hospital-system approved discharge instructions which provide written instruction on how to taper opioid use, links to written/online resources for opioid misuse, overdose prevention, and State-approved disposal options.

INTERVENTIONS:
Behavioral: Life Care Specialist (LCS) — Life Care Specialist (LCS) will :
  * Provide patients with individualized risk assessment for opioid misuse.
  * Act as patient's "Pain Coach." Providing targeted education and behavior-based pain treatment options.
  * Train and provide CWC evidence based non-pharmaceutical pain management techniques, using the Community Resiliency Model.
  * Use the Opioid Risk Tool (ORT) as the method to identity the risk of substance misuse.
  * Provide education, support and resources, as well as local, state, and national resources to enhance the whole health aspect of the position. These resources include but are not limited to: written documents that outline the key concepts of the pain management techniques taught by the LCS and a list of hotlines and websites.
  * LCS, when applicable, will provide education for caretakers on the risk of opioid use and the non -pharmaceutical pain management protocol.
  * Provide follow up for all patients in intervention group.
  Arms: LCS Intervention

SUMMARY:
This is a randomized control trial aimed at learning more about LCS position and the value it provides to the patient's who have sustained upper extremity traumas.

DETAILED DESCRIPTION:
Opioids are psychoactive substances (narcotics) primarily used for pain relief by producing euphoric effects. Although regularly prescribed by physicians, opioids are highly addictive. Examples include, but are not limited to, morphine, codeine, and oxycodone. Opioids block feelings of pain and trigger a release of dopamine. Dependence occurs with repeated use, as the parts of the brain naturally responsible for releasing dopamine rely on the drug for proper function. When avoided, patients can quickly experience severe withdrawal symptoms similar to the flu. In the United States, more than 115 people die from opioid overdose every day. Despite a year-over-year increase in opioid overdose deaths since the year 2000, opioids remain among the most effective medications providers can offer to control pain. Addiction treatment costs near $78.5 billion and rising, less than 10% of people in need receive treatment. Trauma patients are more likely than other types of patients to be under the influence of psychoactive drugs and alcohol use. The strongest risk factor for developing opioid use disorder is pre-existing substance use disorder. Risk factors for opioid overdose mortality include: middle age, history of substance abuse, including prescription and illicit drugs and alcohol, comorbid mental and medical condition, methadone use, unemployment, polysubstance abuse, opioid naivety, sleep apnea, and pain intensity; these are all conditions representative of typical U.S. trauma patient populations. This significant overlap places high importance on implementing alternative solutions to pain management within this population, and aligns with the Center for Disease Control and Prevention, National Conference for Immunization Coalitions and Partnerships (NCICP) research priority alignment to develop and evaluate an innovative prevention strategy to prevent overdose, including those at greatest risk.

According to studies of patients discharged from the hospital after being prescribed a new medication:

* 86% were aware that they had been prescribed new medications.
* Fewer could identify the name (64%) or number (74%) of their new medications of their dosages (56%), the schedule to take them (68%), or the purpose of the prescription (64%.)
* Only 22% could name at least one adverse effect.
* Only 11% could recall being told of any adverse effects.

Orthopaedic surgeons are the third-most frequent providers of opioid prescription medications among physicians, and orthopaedic surgical patients are at the highest risk of chronic postoperative opioid use. Orthopaedic trauma surgeons face a very difficult task in managing acute pain and the consequences associated with over-prescription of opioid analgesics. Most patients with orthopaedic trauma injuries have very painful injuries and need appropriate pain control.

The Christopher Wolf Crusade (CWC) is a non-profit providing preventative solutions, education, and advocacy for the American opioid epidemic. CWC proposes to introduce a Life Care Specialist (LCS) as an integral member of the clinical team, with a focus on "pain coaching" for trauma patients. In an analogous role served by Certified Child Life Specialists (CCLS) in pediatrics, the LCS will introduce orthopaedic trauma patients to non-pharmacologic coping strategies for pain. Further, LCS will provide much needed patient-centric education on individualized risk for opioid misuse, as well as overdose prevention and safe disposal of unused opioids.

This randomized control trial is aimed at learning more about LCS position and the value it provides to the patient's who have sustained upper extremity traumas.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18 years of age or older
* Orthopaedic trauma patients with an isolated upper extremity injury requiring surgery
* Informed consent obtained
* Working cellphone

Exclusion Criteria:

* Enrolled in a study that does not permit co-enrollment
* Unlikely to comply with the follow-up schedule
* Unable to converse, read or write English at elementary school level
* Unlikely to complete surveys at home, access to phone
* Incarcerated
* Pregnant
* Coronavirus Disease 2019 (COVID-19) positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Pain Numerical Rating Scale (NRS) | Day 1, Week 2, Week 6, Month 3
  The NRS is a commonly used pain assessment tool in both clinical practice and research. The NRS asks respondents to rate the intensity of their pain on a scale where "no pain" is scored as 0 and 'the worst pain imaginable" is scored as 10.
Changes in Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance Score | Day 1, Week 2, Week 6, Month 3
  The PROMIS Sleep Disturbance examines respondent's global severity of insomnia, sleep disruption, and sleep quality over the past seven days. Each of the four Likert scale items' raw score are converted to t-scores, ranging from 0 to 100. Like all PROMIS measures, t-scores are normed to the US population, with a mean of 50 and standard deviation of 10. Lower scores indicate better sleep.
Changes in PROMIS Physical Function Score | Day 1, Week 2, Week 6, Month 3
  PROMIS Physical Function measures participants' self-reported capability to conduct physical activity. This includes capturing function in upper extremities and lower extremities (walking or mobility) as well as a respondent's ability to conduct activities of daily living. There are 4-items on the short form questionnaire and respondents report their capabilities to perform each task on a Likert scale from 5, "without any difficulty", to 1, "unable to do". All 4-items' saw scores are summed before being transformed into t-scores ranging from 0 to 100. Higher scores are better and indicate greater physical function.
Changes in PROMIS Pain Interference Score | Day 1, Week 2, Week 6, Month 3
  The PROMIS Pain Interference scale assesses the extent to which pain impedes engagement with social, cognitive, emotional, physical, and recreational activities over the past 7 days. Pain interference is an essential aspect of pain management to capture in order to better understand how pain impacts the activities of individuals rather than subjective severity alone.15 On each of the scale's 4-items respondents choose how much pain impeded a specific function or activity, ranging from 1, "not at all", to 5, "very much". Scores are summed across all items and transformed to a t-score ranging from 0 to 100, with lower t-scores indicate less interference due to pain
Changes in PROMIS Prescription Pain Medication Misuse Score | Day 1, Week 2, Week 6, Month 3
  The PROMIS measure of Prescription Pain Medication Misuse assesses current abuse of prescription pain medication, chiefly opioids. The scale has been validated in patient populations with chronic non-cancer pain and has been found to be highly correlated with the Pain Medication Questionnaire (PMQ).

SECONDARY OUTCOMES:
Inpatient Opioid Utilization | During hospitalization (the average length of stay is 3.16 days)
  Inpatient utilization will be extracted from the electronic health record (EHR) by study staff. Opioid medication dosage will be transformed to a total universal measure known as morphine milligram equivalent (MME). MME will be averaged over the length-of-stay (LOS) for a daily dosage, known as MME/day.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Zelenski, MD, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified outcome data and demographic data will be made available for sharing with other researchers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available for sharing beginning after publication of results from this study and ending July 31 2025.
Access Criteria: Data will be available for sharing with researchers who submit a proposal to the PI and have appropriate Institutional Review Board approval to conduct confirmatory analyses. Data will be shared via Emory approved secure share file transfer service or via Emory's Open Access Dataverse.